CLINICAL TRIAL: NCT01482247
Title: L-Arginine, Vascular Response and Mechanisms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Naomi DL Fisher, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008A052379
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-arginine (Active Comparator)
  Interventions: Dietary Supplement: L-Arginine
- Placebo Supplement (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: L-Arginine — Dietary Supplement
  Arms: L-arginine
Dietary Supplement: Placebo Supplement — Dietary Supplement
  Arms: Placebo Supplement

SUMMARY:
The purpose of the study is to employ the supplement L-arginine to test the hypothesis that activation of blood flow to the brain during cognitive tasks is regulated by nitric oxide in older subjects with diabetes mellitus and/or hypertension (high blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* diabetes and/or hypertension

Exclusion Criteria:

* alzheimers disease, dementia, stroke, active herpes, recent angina or heart attack

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Functional transcranial doppler measures | 6 weeks

SECONDARY OUTCOMES:
Flow Mediated Dilation (FMD) | 6 weeks
Finger Blood Flow - Plethysmography (PAT) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fisher, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States